CLINICAL TRIAL: NCT07093398
Title: A Phase 1 Open-label, Randomised, Crossover Study to Assess the Effect of Food on the Pharmacokinetics (PK) of D3S-001 in Healthy Adult Participants
Brief Title: A Phase 1 Study to Assess Food Effect on the Pharmacokinetics of D3S-001 in Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: D3 Bio (Wuxi) Co., Ltd (Industry)
Collaborators: Fortrea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D3S-001-CP003
Record Dates: First submitted 2025-07-10; First posted 2025-07-30 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Healthy Adult Volunteers
Keywords: D3S-001; D3S-001-CP003; Phase 1; Effect of Food; Healthy Adult Participants

STUDY DESIGN:
Intervention Model Description: This will be a Phase 1, single-centre, open-label, randomised, crossover study in healthy adult male and female participants. Potential participants will be screened within 28 days prior to the first dose. Participants will be admitted into the clinical research unit (CRU) on Day -1 and will be confined until end of study (EOS) or until early termination. On Day 1, participants will be randomised to Group 1 or Group 2. Participants will receive Treatment A or Treatment B in each of 2 periods (Periods 1 and 2; Study Days 1 and 4), once under fasted conditions (Treatment A) and once under fed conditions (Treatment B).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 - Fasted and Fed (Experimental): Period 1 (day 1-3): Treatment A - 600mg D3S-001, following an overnight fast of at least 10 hours.
  Period 2 (day 4 to 6): Treatment B - 600mg D3S-001, administered 30 minutes after the start of a high-fat/high-calorie meal breakfast.
  Interventions: Drug: D3S-001
- Group 2 - Fed and Fasted (Experimental): Period 1 (day 1-3): Treatment B - 600mg D3S-001, administered 30 minutes after the start of a high-fat/high-calorie meal breakfast.
  Period 2 (day 4-6): Treatment A - 600mg D3S-001, following an overnight fast of at least 10 hours.
  Interventions: Drug: D3S-001

INTERVENTIONS:
Drug: D3S-001 — The investigational product dose: 600 mg D3S-001 capsules.
  A 600-mg oral dose of D3S-001 will be given to potential participants on Day 1 and Day 4.

SUMMARY:
The goal of this clinical trial is to Assess the Effect of Food on the

Pharmacokinetics (PK) of D3S-001 in Healthy Adult Participants. The main question[s] it aims to answer are:

1. Evaluate the PK of D3S-001 administered in the fasted and fed state in healthy adult participants.
2. Evaluate the safety and tolerability of D3S-001 administered in the fasted and fed state in healthy adult participants.

Potential participants will be screened within 28 days prior to the first dose. Participants will be admitted into the clinical research unit (CRU) on Day -1 and will be confined until end of study (EOS) or until early termination. On Day 1, participants will be randomised to Group 1 or Group 2. Participants will receive Treatment A or Treatment B in each of 2 periods (Periods 1 and 2; Study Days 1 and 4), once under fasted conditions (Treatment A) and once under fed conditions (Treatment B). Each participant will receive both treatments.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and willing to sign an informed consent form (ICF) and to abide by the study restrictions.
* Males or females of any race, aged between 18 to 65 years, inclusive, with a body mass index between 18.0 and 32.0 kg/m2, inclusive.
* In good health, determined by no clinically significant findings.

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, haematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder.
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance.
* History of stomach or intestinal surgery (including but not limited to cholecystectomy) or resection that would potentially alter absorption and/or excretion of orally administered drugs.
* Unable or unwilling to consume the protocol-specified high-fat breakfast.

Other protocol inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) | From screening to end of treatment at 34 days
  Maximum Observed Concentration (Cmax) of D3S-001 administered in the fasted and fed state.
Area under the concentration-time curve | From screening to end of treatment at 34 days
  Evaluate the area under the concentration-time curve from time zero to the time of the last quantifiable concentration after D3S-001 administered in the fasted and fed state.

SECONDARY OUTCOMES:
Adverse events | From screening to end of study (approximately 34 days)
  Subjects will be observed for any signs or symptoms of adverse events and asked about their condition by open questioning, such as "How have you been feeling since you were last asked?", at least once each day while resident at the study site and at each study visit.
Number of clinically significant clinical laboratory findings | On Screening visit, Day -1, Days 2-3 and Days 5-6 (End of Study)
  Evaluate the safety and tolerability of the drug through clinical laboratory assessments, including clinical chemistry, haematology, coagulation, and urinalysis.
Number of clinically significant electrocardiogram parameters | On screening day, Day -1 and Days 1-6 (End of Study)
  Evaluate the safety and tolerability of the drug using resting 12-lead electrocardiogram (ECG) parameters, recorded after the subject has been supine and at rest for at least 5 minutes. The following ECG Measurements will be recorded: Heart Rate, RR Interval, PR Internal, QRSD QT Interval, QTcB and QTcF.
To determine the safety and tolerability of the drug in healthy subjects, as assessed by the collection of vital signs. | On screening day, Day -1 and Days 1-6 (End of Study)
  Temperature in Degrees Celsius (℃)
To determine the safety and tolerability of the drug in healthy subjects, as assessed by the collection of vital signs. | On screening day, Day -1 and Days 1-6 (End of Study)
  Pulse in beats per minute (bpm)
To determine the safety and tolerability of the drug in healthy subjects, as assessed by the collection of vital signs. | On screening day, Day -1 and Days 1-6 (End of Study)
  Respiratory Rate in respirations per minute (rpm)
To determine the safety and tolerability of the drug in healthy subjects, as assessed by the collection of vital signs. | On screening day, Day -1 and Days 1-6 (End of Study)
  Systolic and Diastolic Blood Pressure in millimeters of mercury (mmHg)
Number of clinically significant physical examinations | On Screening visit, Day -1 and Day 6 (End of Study)
  Evaluate the safety and tolerability of the drug by performing HEENT [head, eyes, ears, nose, and throat], mouth/dental, neck [including thyroid & nodes], cardiovascular, respiratory, gastrointestinal, renal, neurological, musculoskeletal, skin, and other examinations.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Polasek, MD, Principal Investigator — CMAX Clinical Research
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia